CLINICAL TRIAL: NCT04117308
Title: Analysis of the Use of the Fetal Movement Counting for Prolonged Pregnancy: Prospective Randomized Study.
Brief Title: Analysis of the Use of the Fetal Movement Counting for Prolonged Pregnancy.
Acronym: COMPTAMAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18CH201; ANSM (Other: 2019-A00969-48)
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-08

CONDITIONS: Prolonged Pregnancy
Keywords: Perinatal morbidity; Prolonged pregnancy; Fetal active movement count
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized, open-label study evaluating the use of fetal active movements counts on the perinatal morbidity score in patients with prolonged pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients who received a classic information.
  Interventions: Procedure: Classic information
- Educated group (Experimental): Who have been educated to the active fetal movements count.
  Interventions: Procedure: Information by detailed brochure on the fetal active movements account

INTERVENTIONS:
Procedure: Classic information — The team delivers to each patient a unique and standardized information brochure including a definition of fetal active movements, and the need to consult if the patient perceives less the movements of her fetus.
  Arms: Control group
Procedure: Information by detailed brochure on the fetal active movements account — Delayed single and standardized explanatory card on fetal movements (definition, interests of their follow-up, technique of movements on fetuses, table to fill during the follow-up noting the number of active movements physical feelings at 3 times of the day, managing the decrease in the number of active fetal movements).
  Arms: Educated group

SUMMARY:
Prospective mono-centric randomized open-label study (randomization 1: 1, 2 groups) comparing a group of patients who received conventional information to a group of patients who had been sensitized to a fetal active movement count technique.

The study will take place at the University Hospital Center of Saint-Etienne in the gynecology-obstetrics department.

An information brochure on the study will be handed over at the end of the term consultation to 41+0 weeks of gestation. After collecting the consent of the patient, the distribution between the two groups will be done by randomization. Thus, for the fetal active movement count group, fetal active movement count education will be proposed during the term consultation with the submission of an information brochure. The "control" group will also receive a simple information pamphlet with, in writing, what patients currently receive orally: definition of active fetal movements, and the need to consult if the patient perceives less movements of her fetus .The principal objective is to compare perinatal morbidity in relation with the sensation of decrease active fetal movements in case of late pregnancy, according to the fact if the patients use or not the AFM's count.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman presenting herself in the Gynecology-obstetrics Department of the hospital of Saint-Etienne during the term consultation at 41 weeks of amenorrhea + 0 day.
* Non pathological Singleton Pregnancy except for balanced gestational diabetes
* Patient affiliated with or entitled to a Social security plan
* Patients who have given their participation agreement and signing the consent

Exclusion Criteria:

* Woman refusing to participate in the study (lack of consent)
* Non-francophone woman (and / or enable + read french)
* Woman making a maternity change for childbirth (risk of follow-up bias)
* Pathological pregnancy
* Participation to another interventional study.
* Patient subject to legal protection or unable to express consent
* Patient who has already benefited from an awareness of the AFM's account

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
The presence of more than 2 criteria of a composite perinatal morbidity score. | At the delivery.
  The primary outcome will be the presence of more than 2 criteria of a composite perinatal morbidity score:
  * Fetal heart rate anomaly during childbirth.
  * Apgar < 7 at 5 minutes
  * Cord arterial Ph < 7.20
  * Acute respiratory distress with the need for surveillance in neonatal resuscitation

SECONDARY OUTCOMES:
Number of consultations | At the delivery.
  Number of consultations with the sensation of decrease active fetal movements.
Consultation's delay | At the delivery.
  Consultation's delay in relation with the sensation of decrease active fetal movements (classified on <12 hours or >12hours).
Ranking of consultations in 'justified' or 'not justified' | At the delivery.
  Ranking of consultations in 'justified' or 'not justified' is depending on the result of the complementary examinations practiced (Ultrasound with Manning score, kleihauer test). A consultation for reduction of fetal active movements is considered justified if presence of abnormal fetal heart rate and / or Manning score less than 8/8 and / or positive kleihauer test.
Mode of labor | At the delivery.
  Spontaneous or induction of labor, and explications for induction.
Childbirth | At the delivery.
  Caesarean, spontaneous outcome, assisted vaginal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine BARJAT, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No